CLINICAL TRIAL: NCT06918665
Title: HEALTH Trial - Healthy Adult Evaluation of Ivermectin Bioequivalence: Infant Versus Standard Formulation
Acronym: HEALTH
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Difficulty in finalising the intervention
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: Monash University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 118266
Record Dates: First submitted 2025-03-31; First posted 2025-04-09 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-05

CONDITIONS: Scabies
Keywords: ivermectin
MeSH Terms: conditions — Scabies | interventions — Tablets

STUDY DESIGN:
Intervention Model Description: Randomised, Open-Label Cross-over
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (standard 3mg ivermectin tablet then ivermectin infant formula preparation) (Active Comparator): Ivermectin standard 3mg tablet
  washout 21 days
  ivermectin infant formula preparation
  Interventions: Drug: ivermectin infant formula preparation; Drug: Standard ivermectin 3mg tablet
- Sequence 2 (ivermectin infant formula preparation then standard ivermectin 3mg tablet) (Active Comparator): ivermectin infant formula preparation
  21 days washout
  ivermectin standard 3mg tablet
  Interventions: Drug: ivermectin infant formula preparation; Drug: Standard ivermectin 3mg tablet

INTERVENTIONS:
Drug: ivermectin infant formula preparation — The ivermectin infant formula preparation is produced by micronizing the standard 3mg ivermectin tablet and then blending it with Stage 1 infant formula (Blackmores brand) to produce a homogenous powder. This powder blend of ivermectin and infant formula is then filled into food grade clear capsules.
Drug: Standard ivermectin 3mg tablet — standard 3mg ivermectin tablet

SUMMARY:
This is a clinical trial to compare two formulations of the drug ivermectin: the standard 3mg tablet formulation versus a newly developed infant formula preparation. The goal of the trial is to determine if the new formulation functions in the same way, tastes the same and causes no new side effects. The trial will involve 52 participants who will be healthy adult volunteers. The participants will receive both formulations - the order they receive each formulation will be assigned randomly (similar to the toss of a coin).

DETAILED DESCRIPTION:
Randomised open-label cross-over trial of 52 healthy adult volunteers comparing two ivermectin formulations: the standard tablet formulation, and a newly developed infant formula preparation. Participants will be randomised to receive one of these two formulations at the start of the trial and after a 21 day wash out period will be given the alternative formulation. Blood samples will be taken to determine serum drug concentrations. The bioequivalence, tolerability and drug-related adverse effects will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged over 18 years up to 55 years; and
* Body mass index of 18.0 - 32.0 kg/m2 with body weight ≥ 50.0 kg; and
* Medically healthy, determined by medical history, physical examination, no clinically significant abnormalities on baseline blood tests, vital signs (blood pressure, oxygen saturation and heart rate) as deemed by the study Doctor; and
* Females must be non-pregnant, non-lactating or postmenopausal for at least 1 year or surgically sterile for at least 6 months prior to dosing; and
* Sexually active, non-pregnant female participants will be required to use an effective form of contraception from 28 days prior to study until end of study; and
* Males must not have a pregnant partner and must agree to use condoms as a method of contraception from the time of signing informed consent until end of the study; and
* Must be willing and able to read, understand, and sign the participant information and consent form. Willing to comply with all study requirements, including the inpatient period and outpatient visits for the duration of the study; and
* Good venous access on at least one arm as assessed by study staff.

Exclusion Criteria:

* History of any clinically important cardiac, endocrinologic, haematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, and renal, or other major disease, as determined by the study doctor; or
* Known allergy to ivermectin or taking a drug that interacts with ivermectin via the P-glycoprotein transport system (e.g. amiodarone, carvedilol, clarithromycin, clotrimazole); or
* Currently taking warfarin; or
* Known lactose intolerance or cow's protein intolerance; or
* Known elective surgery scheduled within the next 3 months; or
* Inability to comply with the study protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Serum ivermectin Area Under the Curve (AUC) 0-96h bioequivalence across the 2 formulations (standard ivermectin tablet versus new infant formula preparation) | 31 days
  The serum ivermectin Area Under the Curve (AUC) 0-96h for both the new infant formula preparation and the standard 3 mg tablet will be measured. Bioequivalence is defined as the 90% Confidence Interval (CI) of the geometric mean ratio of AUC 0-96h of the infant formula preparation relative to the standard 3mg tablet falling within 80-125%.
Serum ivermectin Maximum Concentration (Cmax) bioequivalence across the 2 formulations (standard ivermectin tablet versus new infant formula preparation) | 31 days
  The serum ivermectin Maximum Concentration (Cmax) for both the new infant formula preparation and the standard 3 mg tablet will be measured. Bioequivalence is defined as the 90% Confidence Interval (CI) of the geometric mean ratio of Cmax of the infant formula preparation relative to the standard 3mg tablet falling within 80-125%.

SECONDARY OUTCOMES:
Safety as measured by the proportion of participants experiencing one or more drug-related adverse effect(s) with each ivermectin formulation | 51 days
  Proportion of participants who experience one or more drug-related adverse effects with each ivermectin formulation
Palatability of the new infant formula preparation as measured by a visual analogue scale (VAS) | 51 days
  Palatability of the new infant formula preparation will be assessed using a visual analogue scale to assess bitterness and overall likeability. The scale used for this VAS tool will be 0 to 10. For the question on overall likeability, a higher score will correspond with a higher level of likeability. For the question on bitterness, a higher score will indicate a higher level of bitterness.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Gwee, Principal Investigator — Murdoch Childrens Research Institute
Locations (1):
- The Royal Children's Hospital, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
Beginning 12 months following analysis and article publication, upon approval of the request, the following will be made available long-term for the use by future researchers from a recognised research institute whose proposed use of the data has been ethically reviewed and approved by an independent committee and who accepts MCRI's condition for access:
  * Individual participant data that underlie the results reported in this article after de-identification (text, tables, figures and appendices)
  * Trial Protocol, PICF

REFERENCES:
- [Background] Hauschke D, Steinijans VW, Pigeot I. Bioequivalence Studies in Drug Development. Chichester: John Wiley; 2007
- [Background] European Medicines Agency. (2010). Guideline on the investigation of bioequivalence (CPMP/EWP/QWP/1401/98 Rev. 1/Corr). Available at https://www.tga.gov.au.
- [Background] Yotsu RR, Fuller LC, Murdoch ME, van Brakel WH, Revankar C, Barogui MYT, Postigo JAR, Dagne DA, Asiedu K, Hay RJ. A global call for action to tackle skin-related neglected tropical diseases (skin NTDs) through integration: An ambitious step change. PLoS Negl Trop Dis. 2023 Jun 15;17(6):e0011357. doi: 10.1371/journal.pntd.0011357. eCollection 2023 Jun. PMID 37319139
- [Background] Engelman D, Marks M, Steer AC, Beshah A, Biswas G, Chosidow O, Coffeng LE, Lardizabal Dofitas B, Enbiale W, Fallah M, Gasimov E, Hopkins A, Jacobson J, Kaldor JM, Ly F, Mackenzie CD, McVernon J, Parnaby M, Rainima-Qaniuci M, Sokana O, Sankara D, Yotsu R, Yajima A, Cantey PT. A framework for scabies control. PLoS Negl Trop Dis. 2021 Sep 2;15(9):e0009661. doi: 10.1371/journal.pntd.0009661. eCollection 2021 Sep. PMID 34473725
- [Background] Ponsonby-Thomas E, Pham AC, Huang S, Salim M, Klein LD, Offersen SM, Thymann T, Boyd BJ. Human milk improves the oral bioavailability of the poorly water-soluble drug clofazimine. Eur J Pharm Biopharm. 2025 Feb;207:114604. doi: 10.1016/j.ejpb.2024.114604. Epub 2024 Dec 13. PMID 39675684
- [Background] Naranjo CA, Busto U, Sellers EM, Sandor P, Ruiz I, Roberts EA, Janecek E, Domecq C, Greenblatt DJ. A method for estimating the probability of adverse drug reactions. Clin Pharmacol Ther. 1981 Aug;30(2):239-45. doi: 10.1038/clpt.1981.154. No abstract available. PMID 7249508
- [Background] Gwee A, Steer A, Phongluxa K, Luangphaxay C, Senggnam K, Philavanh A, Lei A, Martinez A, Huang S, McWhinney B, Ungerer J, Duffull S, Yang W, Zhu X, Coghlan B. Ivermectin therapy for young children with scabies infection: a multicentre phase 2 non-randomized trial. Lancet Reg Health West Pac. 2024 Jul 13;49:101144. doi: 10.1016/j.lanwpc.2024.101144. eCollection 2024 Aug. PMID 39109221
- [Background] Karimkhani C, Colombara DV, Drucker AM, Norton SA, Hay R, Engelman D, Steer A, Whitfeld M, Naghavi M, Dellavalle RP. The global burden of scabies: a cross-sectional analysis from the Global Burden of Disease Study 2015. Lancet Infect Dis. 2017 Dec;17(12):1247-1254. doi: 10.1016/S1473-3099(17)30483-8. Epub 2017 Sep 21. PMID 28941561
- [Background] Dabira ED, Soumare HM, Conteh B, Ceesay F, Ndiath MO, Bradley J, Mohammed N, Kandeh B, Smit MR, Slater H, Peeters Grietens K, Broekhuizen H, Bousema T, Drakeley C, Lindsay SW, Achan J, D'Alessandro U. Mass drug administration of ivermectin and dihydroartemisinin-piperaquine against malaria in settings with high coverage of standard control interventions: a cluster-randomised controlled trial in The Gambia. Lancet Infect Dis. 2022 Apr;22(4):519-528. doi: 10.1016/S1473-3099(21)00557-0. Epub 2021 Dec 15. PMID 34919831